CLINICAL TRIAL: NCT03817567
Title: Phase Ib, Open-label, Single-arm, Multicenter Study to Evaluate Safety and Efficacy of SCT200 in Patients With Advanced Esophageal Squamous Cell Carcinoma Progressed Following Treatment With Taxane/Platinum/Fluorouracil
Brief Title: Safety and Efficacy of SCT200 in Patients With Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT200IbmESCC
Record Dates: First submitted 2019-01-15; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Carcinoma; Carcinoma, Squamous Cell; Esophageal Neoplasms; Neoplasms, Squamous Cell; Esophageal Diseases; Epidermal growth factor receptor; EGFR; SCT200
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Carcinoma; Carcinoma, Squamous Cell; Esophageal Neoplasms; Neoplasms, Squamous Cell; Esophageal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- recombinant anti-EGFR monoclonal antibody（SCT200） (Experimental): 6.0mg/kg QW for 6 weeks, then 8.0mg/kg Q2W
  Interventions: Drug: recombinant anti-EGFR monoclonal antibody

INTERVENTIONS:
Drug: recombinant anti-EGFR monoclonal antibody — Experimental: Recombinant Anti-EGFR Monoclonal Antibody（SCT200）. Initially, SCT200 6.0mg/kg will be administered at day 1 every week for a maximum of 6 cycles. After 6 cycles SCT200 8.0mg/kg will be administered at day 2 every weeks until disease progression.
  Other Names: SCT200

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant anti-EGFR monoclonal antibody（SCT200）in patients with advanced esophageal squamous cell carcinoma progressed following treatment with taxane/platinum/fluorouracil.

DETAILED DESCRIPTION:
This is a open label, single-arm multicenter phase Ib study,and is designed to evaluate Objective Response Rate (ORR) in advanced esophageal squamous cell carcinoma progressed following treatment with taxane/platinum/fluorouracil treated with anti-EGFR monoclonal antibody SCT200.

ELIGIBILITY:
Inclusion Criteria:

* Males or females. Aged 18 to 75 years old;
* Histologically or cytologically proven squamous cell carcinoma of the esophagus, which is locally unresectable or distant metastatic disease;
* Disease progressed following standard therapies. Patients has treated with taxane/platinum/fluorouracil and/or radiotherapy. Failure of standard therapy ：Disease progressed or developed non-tolerable toxicity during or within 3 months after last systemic chemotherapy or radical concurrent chemoradiotherapy. For adjuvant therapy/neoadjuvant therapy, disease relapse or progression during treatment or within 6 months after treatment is considered as failure of standard therapy;
* According to RECIST 1.1 , patients must have at least one measurable lesion which was not treated with local treatment such as radiotherapy. Tumour lesions situated in a previously irradiated area which have been demonstrated progression in the lesion, are considered measurable;
* With an Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* Life expectancy of longer than 3 months ( clinical assessment);
* Adequate organ and marrow function as defined below:

Absolute neutrophil count (ANC) greater than/equal to 1.5×l09/L; Platelets greater than/equal to 75×109/L; Hemoglobin greater than/equal to 80g/L; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than/equal to 3 times ULN, or less than/equal to 5 times ULN if known liver metastases; Total bilirubin less than/equal to 1.5 within institutional limit of normal (ULN); Serum creatinine less than/equal to 1.5 times ULN; Electrolyte: magnesium greater than/equal to normal.

* Women of childbearing potential must not be pregnant as assessed by a negative urine or serum beta HCG test upon admission to the hospital, and must agree to use adequate contraception during the study until to 6 months after the last dose of SCT200.For male,if his sexual partners is child-bearing potential, he should use effective contraception from the time of signing the informed consent form until at least 6 months after the last dose of study drug.
* Able to provide written informed consent and can understand and comply with the requirements of the study;

Exclusion Criteria:

* Patients with active central nervous system metastasis or a history of central nervous system metastasis;(If the subject has been suspected with central nervous system metastasis,imaging examination confirmation must be performed within 28 days to exclude central nervous system metastasis;
* Patients with other primary malignancies except cured of non-melanoma skin cancer, carcinoma in situ of cervix or prostatic intraepithelial neoplasia;
* Patients who are allergic to analogue of SCT200 and/or its inactive ingredients;
* Patients administrated EGFR target treatment including EGFR TKI agent or anti- EGFR monoclonal antibody;
* Within 4 weeks, patients received anti-tumor drugs (such as chemotherapy, hormone therapy, immune therapy, the antibody therapy, radiotherapy) or research drugs, or patients with grade 2 or more adverse reaction caused by previous anti-tumor therapy(except alopecia or neurotoxicity grade 2 or less);
* Patients are currently enrolled in other research devices or in research drugs, or less than 4 weeks from other research drugs or devices;
* Patients received major surgery(such as need general anesthesia ) within 4 weeks , should recover from the injury associated with the surgery;
* Patients treated with EPO, G-CSF or GM-CSF;
* Patients who have clinically significant cardiovascular disease (defined as unstable angina pectoris, symptomatic congestive heart failure (NYHA, greater than II), uncontrollable severe arrhythmia);
* Patients occurred myocardial infarction within 6 months;
* Patients who have interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or CT or MRI reminder ILD ;
* Patients with clinical symptoms, required clinical intervention or stable time less than 4 weeks of serous cavity effusion (such as pleural effusion and ascites);
* Patients with active hepatitis B or active hepatitis C, etc. (for patients with a history of hepatitis B, whether treated or not, HBV DNA ≥104 or ≥ 2000IU/ml, HCV RNA≥15IU/ml); HIV antibody positive (if there is no clinical evidence suggesting that there may be HIV infection, there is no need to detect);
* Patients with uncontrolled active infections before enrollment 2 weeks (except simple urinary tract infection or upper respiratory tract infection);
* Patients have alcohol or drug addiction;
* Patients with serious abnormal medical, psychological or laboratory results history which may affect explanation of study results;
* Subjects are considered not suitable for the study by investigator,who have other conditions that may affect their adherence and the evaluation of study indicators.,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | one year
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment.

SECONDARY OUTCOMES:
Adverse events (AEs) | one year
  AE are assessed according to NCI CTCAE v4.03.
PFS | one year
  PFS is defined as the time from first dose of SCT200 until the date of first documentation of progression or date of death, whichever occurs first,according to RECIST v1.1 criteria.
Duration of response (DOR) | one year
  DOR is defined as time from the date when a patient first meets the criteria for CR or PR according to RECIST v1.1, until the date that progressive disease (PD) is objectively documented or death, whichever occurs first
Overall survival (OS) | one year
  OS is defined as time from first dose of SCT200 until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital., Zhengzhou, Henan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality